CLINICAL TRIAL: NCT01350973
Title: A Phase 3, Multicenter, Double-blind, Parallel-group Study to Evaluate the Efficacy and Safety of TAK-085 in Subjects With Hypertriglyceridemia.
Brief Title: Efficacy of TAK-085 in Participants With Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-085/CCT-002; JapicCTI-090937 (Registry Identifier: JapicCTI); U1111-1120-7801 (Registry Identifier: WHO); JapicCTI-R140452 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Hypertriglyceridemia
Keywords: Drug Therapy
MeSH Terms: conditions — Hypertriglyceridemia | interventions — TAK-085; Omacor; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-085 2 g (Experimental): TAK-085 2 g, orally, once daily for up to 12 weeks.
  Interventions: Drug: Omega-3-acid ethyl esters 90 (TAK-085)
- TAK-085 4 g (Experimental): TAK-085 2 g, orally, twice daily for up to 12 weeks.
  Interventions: Drug: Omega-3-acid ethyl esters 90 (TAK-085)
- EPA-E 1.8 g (Experimental): Eicosapentaenoic acid-ethyl (EPA-E) capsule 0.6 g, orally, three-times daily for up to 12 weeks.
  Interventions: Drug: Eicosapentaenoic acid-ethyl (EPA-E)

INTERVENTIONS:
Drug: Omega-3-acid ethyl esters 90 (TAK-085) — Omega-3-acid ethyl esters 90 (TAK-085) capsules. Each one gram of fatty acid in TAK-085 contains approximately 465 mg of EPA plus 375 mg of docosahexaenoic acid-ethyl as ethyl esters.
  Other Names: LOVAZA; Omacor
  Arms: TAK-085 2 g; TAK-085 4 g
Drug: Eicosapentaenoic acid-ethyl (EPA-E) — EPA-E, 0.6 g, orally, three-times daily for up to 12 weeks.
  Other Names: Atheropan®
  Arms: EPA-E 1.8 g

SUMMARY:
The purpose of this study was to determine the efficacy and safety of TAK-085, once daily (QD) or twice daily (BID), compared to ethyl eicosapentaenoate (EPA-E), three times daily (TID) in participants with hypertriglyceridemia undergoing lifestyle modification.

DETAILED DESCRIPTION:
TAK-085 is an oral capsule medicine licensed to Takeda Pharmaceutical Company Ltd. TAK-085 contains omega-3 fatty acid ethyl (mainly, ethyl eicosapentaenoate (EPA-E) and ethyl docosahexaenoic acid (DHA-E)).

This is a phase 3, double-blind, randomized study to evaluate the efficacy and safety of TAK-085 compared to EPA-E in participants with hypertriglyceridemia who are undergoing lifestyle modification.

The study period is a total of 20 weeks, comprised of an 8- week screening period and 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with values of fasting triglyceride level at Visit 2 (Week -4) and Visit 3 (Week -2) are 150 mg/dL or higher and less than 750 mg/dL, and the difference between these 2 values is within 30% of the higher one.
2. Participants with differences between 2 values of fasting Low density lipoprotein - cholesterol level measured at Visit 2 (Week -4) and Visit 3 (Week -2) are within 25% of the higher one.

Exclusion Criteria:

1. Participants who have coronary artery diseases (eg, confirmed myocardial infarction and angina pectoris) within 6 months prior to Visit 1 (Week -8) or participants with a history of revascularization.
2. Participants who received aortic aneurysmectomy or is complicated with aortic aneurysm within 6 months prior to Visit 1 (Week -8).
3. Participants who have a history or complication of a clinically significant hemorrhagic disease (eg, hemophilia, capillary fragility illness, digestive tract ulcer, urinary tract hemorrhage, hemoptysis, vitreous haemorrhage and so forth) within 6 months prior to Visit 1 (Week -8).
4. Participants who have been diagnosed with pancreatitis.
5. Participants who have been diagnosed with lipoprotein lipase (LPL) deficiency, apolipoprotein C-II deficiency or type III familial hyperlipidemia.
6. Participants with complication of Cushing's syndrome, uremia, systemic lupus erythematosus (SLE) or serum dysproteinemia.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor, Clinical Cell Biology and Medicine, Study Director — Graduate School of Medicine, Chiba University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 69 investigational sites in Japan from 21 November 2009 to 28 December 2010.
Pre-assignment Details: Participants with hypertriglyceridemia were randomized to receive omega-3-acid ethyl esters 90 (TAK-085) 2 g once daily or TAK-085 2 g twice daily or EPA-E 0.6 g three-times daily.
Period: Overall Study
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Started | 206 | 210 | 195
Received Treatment | 205 | 210 | 195
Completed | 200 | 202 | 187
Not Completed | 6 | 8 | 8
Not completed — Adverse Event | 4 | 7 | 7
Not completed — Voluntary Withdrawal | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g | Total
Number analyzed (Participants) | 206 | 210 | 195 | 611
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.76) | 55.0 (10.50) | 55.6 (10.52) | 54.8 (10.60)
Age, Customized [Number; unit: participants]
  ≥20 - <65 years | 168 | 169 | 148 | 485
  ≥65 - ≤74 years | 38 | 41 | 47 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 53 | 38 | 137
  Male | 160 | 157 | 157 | 474
Region of Enrollment [Number; unit: participants]
  Japan | 206 | 210 | 195 | 611
Menopause Status [Number; unit: participants]
  Yes | 36 | 42 | 31 | 109
  No | 8 | 6 | 6 | 20
  Not Applicable | 162 | 162 | 158 | 482
Height, Categorical [Number; unit: participants]
  <160 cm | 49 | 49 | 41 | 139
  ≥160 - <170 cm | 91 | 86 | 78 | 255
  ≥170 cm | 66 | 75 | 76 | 217
Height [Mean (Standard Deviation); unit: cm] | 165.5 (8.60) | 165.7 (8.64) | 166.0 (8.89) | 165.7 (8.69)
Weight, Categorical [Number; unit: participants] — The number of participants with available weight data are 205, 210 and 195 in each treatment arm, respectively.
  participants
    <60.0 kg | 33 | 33 | 33 | 99
    ≥60.0 - <70.0 kg | 58 | 61 | 58 | 177
    ≥70.0 - <80.0 kg | 56 | 68 | 49 | 173
    ≥80.0 kg | 58 | 48 | 55 | 161
Weight [Mean (Standard Deviation); unit: kg] — The number of participants with available weight data are 205, 210 and 195 in each treatment arm, respectively.
  kg | 73.04 (13.139) | 72.20 (12.435) | 72.90 (13.375) | 72.71 (12.962)
Body Mass Index (BMI), Categorical [Number; unit: participants] — The number of participants with available BMI data are 205, 210 and 195 in each treatment arm, respectively.
  participants
    <25.0 kg/m^2 | 75 | 89 | 69 | 233
    ≥25.0 - <30.0 kg/m^2 | 94 | 93 | 99 | 286
    ≥30.0 kg/m^2 | 36 | 28 | 27 | 91
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — The number of participants with available BMI data are 205, 210 and 195 in each treatment arm, respectively.
  kg/m^2 | 26.55 (3.658) | 26.26 (3.846) | 26.34 (3.628) | 26.38 (3.710)
Smoking Classification [Number; unit: participants]
  Never Smoked | 60 | 66 | 54 | 180
  Current Smoker | 78 | 76 | 69 | 223
  Ex-Smoker | 68 | 68 | 72 | 208
Waist Circumference, Categorical [Number; unit: participants] — The number of participants with available waist circumference data are 205, 210 and 195 in each treatment arm, respectively.
  Mean
  participants
    Male <85.0 cm | 23 | 26 | 32 | 81
    Male ≥85.0 cm | 136 | 131 | 125 | 392
    Female <90.0 cm | 25 | 30 | 25 | 80
    Female ≥90.0 cm | 21 | 23 | 13 | 57
Waist Circumference [Mean (Standard Deviation); unit: cm] — The number of participants with available waist circumference data are 205, 210 and 195 in each treatment arm, respectively.
  cm | 91.85 (8.901) | 91.24 (9.376) | 91.51 (9.232) | 91.53 (9.161)
Coronary Artery Disease (CAD) Category [Number; unit: participants] — CAD Patient Categories define the degree of risk of CAD according to Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases. Categories are classified by the degree of risks in the patient [e.g, smoking, hypertension, excluding level of low density lipoprotein cholesterol (LDL-C)]. Category I=Low risk (best), Category II=Middle risk, Category III=High Risk and History of CAD.
  participants
    Category I | 6 | 15 | 4 | 25
    Category II | 95 | 70 | 79 | 244
    Category III | 102 | 124 | 110 | 336
    History of CAD | 3 | 1 | 2 | 6
Hypertension [Number; unit: participants]
  Yes | 123 | 127 | 131 | 381
  No | 83 | 83 | 64 | 230
Diabetes Mellitus (Including Impaired Glucose Tolerance) [Number; unit: participants]
  Yes | 62 | 70 | 67 | 199
  No | 144 | 140 | 128 | 412
Low High Density Lipoprotein - Cholesterol (HDL-C) [Number; unit: participants]
  Yes | 58 | 56 | 60 | 174
  No | 148 | 154 | 135 | 437
Administration of 3-hydroxy 3-methylglutaryl coenzyme A (HMGCoA) Reductase Inhibitor [Number; unit: participants]
  Yes | 89 | 89 | 83 | 261
  No | 117 | 121 | 112 | 350
Triglycerides, Categorical [Number; unit: participants] — The number of participants with available triglyceride data are 205, 210 and 195 in each treatment arm, respectively.
  participants
    <150 mg/dL | 0 | 0 | 1 | 1
    ≥150 - <300 mg/dL | 143 | 146 | 135 | 424
    ≥300 - <500 mg/dL | 59 | 57 | 51 | 167
    ≥500 mg/dL | 3 | 7 | 8 | 18
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — The number of participants with available triglyceride data are 205, 210 and 195 in each treatment arm, respectively.
  mg/dL | 269.0 (77.52) | 277.5 (97.29) | 271.8 (91.53) | 272.8 (89.12)
Low Density Lipoprotein - Cholesterol (LDL-C), Categorical [Number; unit: participants] — The number of participants with available LDL-C data are 205, 210 and 195 in each treatment arm, respectively.
  participants
    <140 mg/dL | 140 | 149 | 124 | 413
    ≥140 mg/dL | 65 | 61 | 71 | 197
Low Density Lipoprotein - Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — The number of participants with available LDL-C data are 205, 210 and 195 in each treatment arm, respectively.
  mg/dL | 127.4 (29.08) | 125.7 (28.50) | 130.1 (30.54) | 127.7 (29.37)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Triglyceride Level at the Final Visit
Description: The percentage change between triglycerides collected at the end of study drug administration (the end of treatment period or discontinuation) relative to Baseline. Analysis of Covariance (ANCOVA) model was employed, using the Baseline triglyceride level as covariate and the treatment group as an independent variable.
Time Frame: Baseline and 12 weeks
Population: Full analysis set including all participants who were randomized and received at least one dose of the investigational product and with available data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 203 | 208 | 194
percent change | -10.93 (1.6434) [-14.1610 to -7.7062] | -22.65 (1.6238) [-25.8436 to -19.4655] | -11.30 (1.6807) [-14.6014 to -7.9998]
Statistical Analysis 1: Comparison: TAK-085 2 g vs EPA-E 1.8 g; Test type: Superiority or Other; p = 0.8760, ANCOVA — An ANCOVA model was employed, using the baseline triglyceride level as covariate and the treatment group as an independent variable; LS Mean Difference = 0.37, 95% CI 2-sided [-4.2491 to 4.9830]
Statistical Analysis 2: Comparison: TAK-085 4 g vs EPA-E 1.8 g; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -11.35, 95% CI 2-sided [-15.9442 to -6.7637]

2. Secondary Outcome: Percent Change From Baseline in Triglyceride Level Over Time
Description: The percentage change between triglycerides collected at each study visit relative to Baseline.
Time Frame: Baseline and Weeks 4, 8, 10 and 12
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
percent change
  Week 4 (n=203, 208, 192) | -13.085 (26.4479) | -26.939 (20.9540) | -11.417 (27.8599)
  Week 8 (n=199, 205, 191) | -12.055 (23.5955) | -22.501 (29.7039) | -11.321 (29.6792)
  Week 10 (n=198, 202, 188) | -9.707 (25.9148) | -23.436 (31.7008) | -11.416 (28.4762)
  Week 12 (n=198, 199, 185) | -11.707 (27.6764) | -22.606 (25.1665) | -12.431 (31.0903)

3. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein - Cholesterol (LDL-C) Level Over Time
Description: The percentage change between low-density lipoprotein cholesterol collected at each study visit relative to Baseline. Low-density lipoprotein cholesterol particles measured directly by nuclear magnetic resonance.
Time Frame: Baseline and Weeks 4, 8, 10 and 12
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
percent change
  Week 4 (n=203, 208, 194) | 1.120 (16.0172) | 2.262 (15.5408) | -3.409 (13.5003)
  Week 8 (n=200, 205, 191) | -0.846 (15.5473) | -0.420 (17.7696) | -3.008 (13.8462)
  Week 10 (n=199, 202, 188) | -3.055 (15.6128) | -0.862 (18.0310) | -4.297 (14.0827)
  Week 12 (n=199, 200, 187) | -1.639 (16.3582) | -1.056 (18.2732) | -3.393 (17.2972)

4. Secondary Outcome: Percent Change From Baseline in Total Cholesterol Over Time
Description: The percentage change between total cholesterol measured at each study visit relative to Baseline.
Time Frame: Baseline and Weeks 4, 8, 10 and 12
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
percent change
  Week 4 (n=203, 208, 194) | -0.841 (10.0601) | -2.707 (9.0969) | -3.152 (8.1026)
  Week 8 (n=200, 205, 191) | -1.996 (9.5190) | -2.887 (9.7964) | -3.097 (9.2770)
  Week 10 (n=199, 202, 188) | -3.054 (9.0927) | -3.949 (10.5345) | -4.355 (9.1420)
  Week 12 (n=199, 200, 187) | -2.649 (9.4133) | -3.243 (10.6025) | -3.880 (10.8594)

5. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein - Cholesterol (HDL-C) Level Over Time
Description: The percentage change between high-density lipoprotein cholesterol collected at each study visit relative to Baseline.
Time Frame: Baseline and Weeks 4, 8, 10 and 12
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
percent change
  Week 4 (n=203, 208, 194) | 2.990 (10.5365) | 4.075 (10.9735) | 0.934 (11.6203)
  Week 8 (n=200, 205, 191) | 1.547 (11.6333) | 3.936 (12.4198) | 1.826 (10.1747)
  Week 10 (n=199, 202, 188) | 2.258 (10.6907) | 4.219 (12.0895) | 1.860 (11.0573)
  Week 12 (n=199, 200, 187) | 2.685 (10.8647) | 4.564 (12.7497) | 1.741 (10.8185)

6. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein - Cholesterol Level Over Time
Description: The percentage change between non-high-density lipoprotein cholesterol collected at each study visit relative to Baseline. Non-high-density lipoprotein cholesterol calculated by subtracting high-density lipoprotein cholesterol from total cholesterol.
Time Frame: Baseline and Weeks 4, 8, 10 and 12
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
percent change
  Week 4 (n=203, 208, 194) | -1.955 (12.7395) | -4.634 (11.3386) | -4.274 (10.8403)
  Week 8 (n=200, 205, 191) | -3.022 (11.2524) | -4.931 (11.9003) | -4.418 (11.5415)
  Week 10 (n=199, 202, 188) | -4.624 (11.2058) | -6.190 (12.9755) | -5.994 (11.1866)
  Week 12 (n=199, 200, 187) | -4.159 (11.5205) | -5.384 (13.2602) | -5.140 (14.3444)

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Time Frame: 12 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
participants | 88 | 76 | 83

8. Secondary Outcome: Number of Participants With TEAEs Associated With Abnormal Changes in Vital Signs
Time Frame: 12 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
participants | 1 (10.81) | 0 (10.61) | 0 (10.92)

9. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Chemistry, Hematology or Urinalysis
Time Frame: 12 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
participants | 11 | 11 | 7

10. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings After Study Drug Administration
Time Frame: 12 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 205 | 210 | 195
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Collection of AEs commenced from the time that the subject was first administered investigational product (Week 0). Routine collection of AEs continued until the completion of study treatment (12 weeks of administration)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Serious Adverse Events (participants affected / at risk) | 1/205 | 4/210 | 2/195
Other Adverse Events (participants affected / at risk) | 22/205 | 9/210 | 20/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-085 2 g (N=205) | TAK-085 4 g (N=210) | EPA-E 1.8 g (N=195)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-085 2 g (N=205) | TAK-085 4 g (N=210) | EPA-E 1.8 g (N=195)
Nasopharyngitis (Infections and infestations) | 22 | 9 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.